CLINICAL TRIAL: NCT02867332
Title: A Dose-escalation Phase I Trial of PD-1 Knockout Engineered T Cells for the Treatment of Metastatic Renal Cell Carcinoma
Brief Title: PD-1 Knockout Engineered T Cells for Metastatic Renal Cell Carcinoma.
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No funding
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Wujiang Liu, Professor, Peking University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11007965940
Record Dates: First submitted 2016-08-11; First posted 2016-08-15 (Estimated); Last update posted 2019-03-06 (Actual); Status verified 2016-08

CONDITIONS: Metastatic Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Cyclophosphamide; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test group (Experimental): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will be knocked out by CRISPR Cas9 in the laboratory (PD-1 Knockout T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion. A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third.Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/ day (if tolerant). Patients will receive a total of 2, 3, 4 cycles of treatment.
  Interventions: Biological: PD-1 Knockout T Cells; Drug: Cyclophosphamide; Drug: IL-2
- Comparable group (Placebo Comparator): Peripheral blood lymphocytes will be collected and Programmed cell death protein 1(PDCD1) gene will not be knocked out by CRISPR Cas9 in the laboratory (PD-1 Wild-type T cells). The lymphocytes will be selected and expanded ex vivo and infused back into patients. Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  A total of 2 x 10^7/kg PD-1 Knockout T cells will be infused in one cycle. Each cycle is divided into three administrations, with 20% infused in the first administration, 30% in the second, and the remaining 50% in the third.Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/ day (if tolerant). Patients will receive a total of 2, 3, 4 cycles of treatment.
  Interventions: Drug: Cyclophosphamide; Drug: IL-2

INTERVENTIONS:
Biological: PD-1 Knockout T Cells — PD-1 Knockout T Cells and PD-1 wild-type T Cells will be made by Cell Biotech Co., Ltd. 2x107/kg T cells will be used for test group and comparable group separately.
  Arms: Test group
Drug: Cyclophosphamide — Cyclophosphamide at 20mg/kg single dose will be administered 3 days i.v. before cell infusion.
  Interleukin-2 (IL-2) will be given in the following 5 days, 720000 international unit（IU）/Kg/day (if tolerant).
  Other Names: cytophosphane
Drug: IL-2 — Interleukin-2 (IL-2) will be given in the following 5 days after cell infusion, 720000 international unit（IU）/Kg/ day (if tolerant).
  Other Names: Interleukin-2 (IL-2)

SUMMARY:
This study will evaluate the safety of PD-1 knockout engineered T cells in treating metastatic advanced renal cancer. Blood samples will also be collected for research purposes.

DETAILED DESCRIPTION:
This is a dose-escalation study of ex-vivo knocked-out, expanded, and selected PD-1 knockout-T cells from autologous origin. Patients are assigned to 1 of 3 treatment groups to determine the maximal tolerant dose. After the lower number of cycles are considered tolerant, an arm of the next higher number of cycles will be open to next patients. Biomarkers and immunological markers are collected and analyzed as well.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically verified stage IV Renal cancer with measurable lesions (On CT: longest diameter of tumoral lesion >=10 mm, shorted diameter of lymph node >=15 mm; measurable lesions should not have been irradiated)
* Progressed after all standard treatment
* Performance score: 0-1
* Expected life span: >= 6 months
* Toxicities from prior treatment has resolved. Washout period is 4 weeks for chemotherapy, and 2 weeks for targeted therapy
* Major organs function normally
* Women at pregnant ages should be under contraception
* Willing and able to provide informed consent

Exclusion Criteria:

* Pathology is mixed type
* Emergent treatment of tumor emergency is needed
* Poor vasculature
* Coagulopathy, or ongoing thrombolytics and/or anticoagulation
* Blood-borne infectious disease, e.g. hepatitis B
* History of mandatory custody because of psychosis or other psychological disease inappropriate for treatment deemed by treating physician
* With other immune diseases, or chronic use of immunosuppressants or steroids
* Compliance cannot be expected
* Other conditions requiring exclusion deemed by physician

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11; Primary Completion 2020-11 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events and/or Dose Limiting Toxicities as a Measure of Safety and tolerability of dose of PD-1 Knockout T cells using Common Terminology Criteria for Adverse Events (CTCAE v4.0) in patients | Dose Escalation - Approximately 6 months

SECONDARY OUTCOMES:
Response Rate:Response will be evaluated according to RECIST v1.1 | 90 days
Progression free survival - PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to average 10 months
Overall Survival - OS | The time from randomization to death from any cause, assessed up to 2 years
Peripheral blood circulating tumor DNA | 6 weeks
Temporal Interleukin-2 change in the peripheral blood | Baseline and 1 month and 3 months
Temporal Interferon-γ change in the peripheral blood | Baseline and 1 month and 3 months
Temporal Interleukin-6 change in the peripheral blood | Baseline and 1 month and 3 months

IPD SHARING:
Plan to Share IPD: Undecided
plan to do

REFERENCES:
- [Background] Gandini S, Massi D, Mandala M. PD-L1 expression in cancer patients receiving anti PD-1/PD-L1 antibodies: A systematic review and meta-analysis. Crit Rev Oncol Hematol. 2016 Apr;100:88-98. doi: 10.1016/j.critrevonc.2016.02.001. Epub 2016 Feb 10. PMID 26895815
- [Result] Koshkin VS, Rini BI. Emerging therapeutics in refractory renal cell carcinoma. Expert Opin Pharmacother. 2016 Jun;17(9):1225-32. doi: 10.1080/14656566.2016.1182987. Epub 2016 May 23. PMID 27112171
- [Result] Hofmann L, Forschner A, Loquai C, Goldinger SM, Zimmer L, Ugurel S, Schmidgen MI, Gutzmer R, Utikal JS, Goppner D, Hassel JC, Meier F, Tietze JK, Thomas I, Weishaupt C, Leverkus M, Wahl R, Dietrich U, Garbe C, Kirchberger MC, Eigentler T, Berking C, Gesierich A, Krackhardt AM, Schadendorf D, Schuler G, Dummer R, Heinzerling LM. Cutaneous, gastrointestinal, hepatic, endocrine, and renal side-effects of anti-PD-1 therapy. Eur J Cancer. 2016 Jun;60:190-209. doi: 10.1016/j.ejca.2016.02.025. Epub 2016 Apr 13. PMID 27085692
- [Result] Gunturi A, McDermott DF. Potential of new therapies like anti-PD1 in kidney cancer. Curr Treat Options Oncol. 2014 Mar;15(1):137-46. doi: 10.1007/s11864-013-0268-y. PMID 24504486
- [Result] Bockorny B, Dasanu CA. Intrinsic immune alterations in renal cell carcinoma and emerging immunotherapeutic approaches. Expert Opin Biol Ther. 2013 Jun;13(6):911-25. doi: 10.1517/14712598.2013.778970. Epub 2013 Apr 16. PMID 23586712
- [Derived] Yi L, Li J. CRISPR-Cas9 therapeutics in cancer: promising strategies and present challenges. Biochim Biophys Acta. 2016 Dec;1866(2):197-207. doi: 10.1016/j.bbcan.2016.09.002. Epub 2016 Sep 15. PMID 27641687